CLINICAL TRIAL: NCT00965289
Title: Front-line High-dose Chemotherapy (HDT) Combined With Rituximab for Adults With Aggressive Large B-cell Lymphoma (DLBCL) : Goelams 074 Trial.
Brief Title: High-dose Chemotherapy With Rituximab for Adults With Aggressive Large B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: French Innovative Leukemia Organisation (Other); Hoffmann-La Roche (Industry)
Responsible Party: Pr Noel MILPIED, NANTES UNIVERSITY HOSPITAL /GOELAMS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOELAMS 074
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: B-Cell Lymphoma
Keywords: Aggressive large B-cell lymphoma (DLBCL); Intensive chemotherapy; Rituximab; ASCT
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HDT combined with rituximab before ASCT (Experimental): The study treatment consisted on 2 courses of high-dose R-CHOP-like regimen, followed by a course of high-dose methotrexate with cytarabin. For patients who achieved at least a PR, ASCT started with a BEAM regimen.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab infusion on day 1 dose: 375mg/m²
  Other Names: Mabthera®

SUMMARY:
A prospective pilot trial was proposed to patients with DLBCL, with IH or high adjusted IPI, up to the age of 60 y.o. This program consisted of 2 courses of high-dose R-CHOP-like regimen, followed by a course of high-dose methotrexate with cytarabin. For patients who achieved at least a PR, ASCT started with a BEAM regimen.

DETAILED DESCRIPTION:
Superiority of HDT with autologous stem cell transplantation (ASCT) in the upfront treatment of poor-risk DLBCL remains an option for intermediate-high (IH) or high IPI young adults. We updated results of the prospective trial Goelams 074 to evaluate long-term efficacy and toxicity in 42 patients who underwent HDT with ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 y.o
* Aggressive Large B-Cell Lymphoma (CD20+)
* Ann Arbor stage III, IV
* IH or high adjusted IPI
* signed inform consent

Exclusion Criteria:

* Age < 18 ou > 60 y.o
* other type of lymphoma
* serology VIH +
* other neoplasms apart from basal cell carcinoma or situ carcinoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2002-04; Primary Completion 2003-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
CR rate after 3 high dose chemotherapy courses | safety/efficacy of chemotherapy treatment

SECONDARY OUTCOMES:
CR and PR rate at the end of the study treatment | safety/efficacy of treatment30 days after the end of post ASCT aplasia
PFS,EFS and OS | safety/efficacy of study treatment
Tolerance of Rituximab combined with chemotherapy | safety/efficacy of immunotherapy combined with chemotherapy treatment

CONTACTS AND LOCATIONS:
Overall Officials: Noel MILPIED, PD MS, Principal Investigator — CHU NANTES/GOELAMS
Locations (1):
- University Hospital, Nantes, France